CLINICAL TRIAL: NCT06743581
Title: Phase I/II Study of Combined Treatment With Cemiplimab (Anti-PD-1) and Dupilumab (Anti-IL-4R) in Patients With Early-stage, Resectable NSCLC
Brief Title: Phase I/II Study of Neoadjuvant Cemiplimab and Dupilumab in Early-Stage Non-Small Cell Lung Cancer
Acronym: Dupi-Cemi
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-12543
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Non-Small Cell Lung Cancer; Immunotherapy; Neoadjuvant Therapy
Keywords: NSCLC; Neoadjuvant immunotherapy; Cemiplimab; Dupilumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab; dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant cemiplimab and dupilumab combination therapy (Experimental): Neoadjuvant immunotherapy administered prior to thoracic surgery
  Interventions: Drug: Cemiplimab; Drug: Dupilumab

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab 350 mg administered intravenously on day 1
Drug: Dupilumab — Dupilumab 600 mg administered subcutaneously on day 1

SUMMARY:
This phase 1b/2a study evaluates the safety, feasibility, and efficacy of combining dupilumab (anti-IL-4Rα) and cemiplimab (anti-PD-1) in patients with early-stage, resectable NSCLC. Phase 1b focuses on safety and feasibility, using a 3+3 design to monitor dose-limiting toxicities (DLTs), while Phase 2a assesses the major pathological response (MPR) rate with a Simon's two-stage minimax design. Secondary endpoints include event-free survival, overall survival, and translational objectives such as deep immune monitoring from patient samples, with the trial expected to enroll 24 patients at CHUM over five years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of NSCLC is required before treatment (however, patients with a smoking history and radiographic findings suggestive of NSCLC may consent prior to biopsy to combine research and diagnostic procedures.
* Age ≥ 18 years.
* ECOG performance status 0-1
* Determined to be a surgical candidate for tumor resection by a multidisciplinary team.
* Women of childbearing potential and men must use approved contraception during the study and for 4 months post-treatment. Pregnancy or suspected pregnancy must be reported immediately.
* Adequate organ and marrow function.
* Pre-treatment biopsies are mandatory, and tumors must be T1b or larger (>1cm) and amenable to biopsy as determined by a multidisciplinary team.
* Patients must consent to provide blood at designated study time points.
* Patients must consent to core needle biopsies (at least 3 samples, as deemed safe by the performing surgeon/radiologist) prior to treatment initiation

Exclusion Criteria:

* History of autoimmune disorders or use of immunomodulatory drugs (including dupilumab) within 2 months prior to treatment initiation.
* Active autoimmune disease requiring systemic treatment in the past year, excluding replacement therapies like thyroxine or insulin.
* Use of immunosuppressive drugs or systemic steroids within 7 days prior to treatment, except chronic steroids ≤10mg prednisone or equivalent.
* No smoking history or confirmed tissue or ctDNA evidence of actionable driver alterations (e.g. EGFR mutation, ALK, or ROS1 rearrangements)
* Prior chemotherapy or radiotherapy for another primary tumor, or prior locoregional therapy to the target lesion. Therapy for a different cancer is acceptable.
* Metastatic disease where surgery would not have curative intent.
* Uncontrolled illness, including active infections requiring antibiotics, symptomatic heart failure, unstable angina, or psychiatric/social conditions impeding study compliance.
* Pregnancy or nursing, due to potential harm to the fetus or infant.
* Progressive malignancy requiring active treatment, except for certain stable cancers treated with curative intent
* HIV infection with detectable viral load or not on a stable HAART regimen
* Active Hepatitis B or C (PCR-detectable)
* History of allogeneic hematopoietic or solid organ transplantation.
* Documented hypersensitivity to protein therapeutics.
* Any condition, therapy, or abnormality that may interfere with trial results, patient participation, or their best interest as per the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Safety | First 30 days after immunotherapy
  (Phase 1b) Determine the safety (dose-limiting toxicities) of combined treatment with anti-IL-4R-alpha (dupilumab) and anti-PD-1 (cemiplimab) in patients with early-stage, resectable NSCLC.
Major pathological response (MPR) rate | Day of surgery
  (Phase 2a) Assess efficacy of combined cemiplimab and dupilumab in patients with early stage, resectable NSCLC. Efficacy is defined as percentage of patients achieving major pathological response (MPR), i.e. 90% or greater tumor necrosis at time of resection.

SECONDARY OUTCOMES:
Rate of curative-intent surgery | Day of surgery
  (Phase 1b and 2a) Describe and quantify rate of curative-intent surgery following treatment intervention
Tolerability | For up to 5 years or until death
  (Phase 2a) Assess general tolerability in patients treated with dupilumab and cemiplimab treatment combination
Event-free survival (EFS) | For up to 5 years or until death
  (Phase 1b and 2a) Assess event free survival (EFS) as it relates to neoadjuvant cemiplimab and dupilumab treatment combination and following surgery
Overall survival (OS) | For up to 5 years or until death
  (Phase 1b and 2a) Assess overall survival (OS) as it relates to dupilumab and cemiplimab treatment combination and following surgery
Pathological complete response (pCR) rate | Day of surgery
  (Phase 1b and 2a) Assess pathological complete response (pCR) rate

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Desilets, MD, MSc, Principal Investigator — CHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] LaMarche NM, Hegde S, Park MD, Maier BB, Troncoso L, Le Berichel J, Hamon P, Belabed M, Mattiuz R, Hennequin C, Chin T, Reid AM, Reyes-Torres I, Nemeth E, Zhang R, Olson OC, Doroshow DB, Rohs NC, Gomez JE, Veluswamy R, Hall N, Venturini N, Ginhoux F, Liu Z, Buckup M, Figueiredo I, Roudko V, Miyake K, Karasuyama H, Gonzalez-Kozlova E, Gnjatic S, Passegue E, Kim-Schulze S, Brown BD, Hirsch FR, Kim BS, Marron TU, Merad M. An IL-4 signalling axis in bone marrow drives pro-tumorigenic myelopoiesis. Nature. 2024 Jan;625(7993):166-174. doi: 10.1038/s41586-023-06797-9. Epub 2023 Dec 6. PMID 38057662